CLINICAL TRIAL: NCT00641433
Title: Topical Collagen-Silver Versus Standard Care Following Phenol Ablation of Ingrown Nails: A Randomized Controlled Trial
Brief Title: Topical Collagen-Silver Versus Standard Care Following Removal of Ingrown Nails
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Responsible Party: Office of Sponsored Research, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORT 014
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Ingrown Nail
Keywords: chemocautery
MeSH Terms: conditions — Nails, Ingrown | interventions — Silver Sulfadiazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental (Experimental): Subjects will daily dress their nail bed with oxidized regenerated cellulose collagen-silver, until healing occurs.
  Interventions: Device: oxidized regenerated cellulose collagen-silver
- Control (Active Comparator): Topical silver sulfadiazine cream will be applied daily to the wound bed until healing has occured.
  Interventions: Drug: topical silver sulfadiazine cream

INTERVENTIONS:
Device: oxidized regenerated cellulose collagen-silver — Wound dressed daily with oxidized regenerated cellulose collagen-silver matrix.
  Other Names: Prisma
  Arms: experimental
Drug: topical silver sulfadiazine cream — Cream will be applied to nailbed daily and dressed with a bandage until healing occurs.
  Other Names: Silvadene, Thermazene
  Arms: Control

SUMMARY:
This study's purpose is to prospectively determine whether topical therapy with an oxidized regenerated cellulose collagen-silver compound is more effective than the current standard of topical antibiotic therapy for care following the removal of an ingrown toenail. Eighty adult patients with ingrown toenails will be recruited. Each patient will randomly be assigned to apply either topical silver sulfadiazine cream (standard antibiotic) or the novel collagen-silver compound to their nail bed daily, following removal of the ingrown portion of nail. Patients will return for follow up visits weekly, until healing has occurred or twelve weeks have passed. Healing will be defined as resolution of drainage and inflammatory changes surrounding the nail border.

ELIGIBILITY:
Inclusion Criteria:

* Ingrown toenails will be defined as any incurvated nail border that digs into the skin of the nail fold and causes pain and discomfort

Exclusion Criteria:

* Patients with immunocompromised states

  * chronic steroid use
  * diabetes mellitus
  * collagen vascular disease
  * HIV infection
* Cellulitis proximal to the hallux interphalangeal joint or peripheral vascular disease will be excluded
* We will define peripheral vascular disease as the absence of one or more pedal pulses or the presence of dystrophic changes to the integument

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-11; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
time to healing | weekly

SECONDARY OUTCOMES:
time to return to regular shoe gear | weekly
days unable to work | weekly

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM, PhD, Principal Investigator — Rosalind Franklin University
Locations (2):
- United States (2):
  - Scholl Foot and Ankle Center, North Chicago, Illinois
  - Preofessional Education and Research Institutue, Roanoke, Virginia